CLINICAL TRIAL: NCT07174206
Title: FAPO-2: Cardiac Patient Monitoring Tool for Clinical Observation and Arrhythmia Detection
Acronym: FAPO-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Samsung Eletrônica da Amazônia Ltda (Unknown)
Responsible Party: Principal Investigator, Fabio Biscegli Jatene, Full Professor of Cardiovascular Surgery at the University of São Paulo Medical School (FMUSP) and General Director of InCor-HCFMUSP, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 80963624.2.0000.0068
Record Dates: First submitted 2025-08-19; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Heart Diseases; Atrial Fibrillation (AF); Angina, Unstable
Keywords: Atrial Fibrillation; FAPO; PAOF; Telemonitoring; Digital Health; Arrhythmias
MeSH Terms: conditions — Heart Diseases; Atrial Fibrillation; Angina, Unstable; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: FAPO-2 adopts a prospective, single-group interventional study model in which all participants are remotely monitored using both the smartwatch and a portable holter system. The intervention consists of a structured teleconsultation model triggered by predefined clinical thresholds and critical patterns identified through continuous data integration on the FAPO-SI³ platform. Physiological and biometric data are collected viaHealth applications and transmitted daily (D+1) to the clinical team for near-real-time review. Upon detection of critical events or out-of-range parameters, the system automatically generates alerts that prompt nurse- or physician-led teleconsultations. During these teleconsultations, patient symptoms are evaluated, medication regimens may be adjusted, and decisions are made regarding the need for in-person clinical evaluation.
Who Masked: Outcomes Assessor
Masking Description: ECG Reader: The ECG reader will analyze the ECGs without access to identifiable participant information, ensuring that the interpretation of data is done blindly, without bias related to the patient's identity.
  AI Model Developer: The developer will also work with anonymized data, meaning they will not have access to personal information of the participants, ensuring the integrity and confidentiality of the data during model development.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pilot Group (Experimental): Healthy volunteers monitored for ~14±3 days using both a smartwatch and a portable holter system to validate usability, skin tolerability, signal integrity, and data flow within the platform.
  Interventions: Device: Smartwatch - all data; Device: Portable holter system; Procedure: Telemonitoring; Other: AI Model Development
- Extensive Ambulatory Monitoring Group (Active Comparator): Patients with chronic cardiovascular diseases monitored over 45±3 days. For 30 days, participants use the smartwatch to collect blood pressure, oxygen saturation (SpO2), heart rate (HR), and sigle-lead ECG. Also, for 15 days, participants use both smartwatch (HR and ECG only) and portable holter system simultaneously, with the patch providing continuous ECG monitoring.
  Interventions: Device: Smartwatch - all data; Device: Portable holter system; Procedure: Telemonitoring; Other: AI Model Development
- Extensive Post-Intervention Monitoring (Active Comparator): Patients who have recently undergone minimally invasive cardiovascular procedures such as angioplasty, transcatheter aortic valve implantation (TAVI), or catheter ablation. Monitoring occurs over 45±3 days. For 30 days, participants use the smartwatch to collect blood pressure, oxygen saturation (SpO2), heart rate (HR), and single-lead ECG. Also, for 15 days, both the smartwatch (HR and ECG only) and the portable holter system are used simultaneously, with the portable holter system providing continuous ECG monitoring.
  Interventions: Device: Smartwatch - all data; Device: Portable holter system; Procedure: Telemonitoring; Other: AI Model Development
- Optimized Outpatient Monitoring (Active Comparator): Patients with stable chronic cardiac disease monitored for 15±3 days using both the smartwatch captures heart rate and single-lead ECG, while the portable holter system provides continuous ECG monitoring.
  Interventions: Device: Portable holter system; Procedure: Telemonitoring; Other: AI Model Development; Device: Smartwatch - ECG and HR

INTERVENTIONS:
Device: Smartwatch - all data — Single-lead ECG, blood pressure (BP), oxygen saturation (SpO2), and continuous heart rate (HR).
  Arms: Extensive Ambulatory Monitoring Group; Extensive Post-Intervention Monitoring; Pilot Group
Device: Portable holter system — continuous ECG monitoring for 14 days for comparison with the data from the smartwatch
Procedure: Telemonitoring — Remote consultations triggered by critical alerts based on predefined thresholds.
Other: AI Model Development — Data analysis using artificial intelligence for prioritization of patients based on health data collected from wearables.
Device: Smartwatch - ECG and HR — Single-lead ECG and continuous heart rate (HR)
  Arms: Optimized Outpatient Monitoring

SUMMARY:
The FAPO-2 study (Patient Monitoring Tool for Clinical Observation and Arrhythmia Detection) is a prospective, interventional, non-randomized study designed to evaluate the feasibility, usability, clinical effectiveness, and cost-efficiency of a wearable-enabled remote monitoring strategy in adult cardiac patients. The intervention consists of active clinical management of patients via teleconsultations, triggered by automated alerts generated through wearable data integrated into a centralized digital platform. FAPO-2 will include patients with chronic cardiovascular conditions and those undergoing recent minimally invasive interventions. The central objective is to validate a structured model for early arrhythmia detection, remote risk stratification, and timely clinical action. A total of 520 patients aged ≥22 years will be enrolled, stratified by sex (1:1), and followed at the Heart Institute (InCor) of the University of São Paulo. Participants will be allocated into one of four protocol groups:

Group 1 - Pilot (n=15): Healthy volunteers monitored for ~14±3 days using both the smartwatch and a portable holter system to validate usability, skin tolerability, signal integrity, and data flow within the platform.

Group 2 - Extensive Outpatient Monitoring (n=150): Patients with chronic cardiovascular diseases monitored over a 45-day period. During 30 days, monitoring will be performed using a smartwatch to capture blood pressure, oxygen saturation, heart rate, and single-lead ECG. For 15 days, participants will use both the smartwatch (for HR and ECG) and a portable holter system.

Group 3 - Extensive Post-Intervention Monitoring (n=50): Patients recently undergoing procedures such as angioplasty, TAVI, or ablation, following the same monitoring protocol as Group 2.

Group 4 - Optimized Outpatient Monitoring (n=305): Patients with stable chronic cardiac disease monitored for 15±3 days, using both devices simultaneously for HR and ECG (smartwatch) and portable holter system.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cardiovascular disease, of both sexes, aged over 22 years;
* Provision of informed consent through signature of the Informed Consent Form (ICF);
* Assentation to adhere to study procedures and requirements;
* Patients indicated for outpatient follow-up due to a cardiovascular condition, or with clinical parameters indicating the need for conventional surgical or catheter-based interventions (e.g., catheter ablation for arrhythmias, transcatheter aortic valve implantation, percutaneous coronary intervention, etc.);
* Low or no risk of skin injury, based on Braden Scale clinical criteria or clinical team assessment

Exclusion Criteria:

* Presence of skin conditions, such as vitiligo, lupus, or atopic dermatitis, as well as tattoos on the wrist that may interfere with the smartwatch's optical sensor readings;
* Known sensitivity or history of allergic reactions to components of the wearable devices or related items, such as adhesives or electrodes;
* Inability to properly use the wearable monitoring devices due to physical, cognitive, or technological limitations;
* Presence of a peripherally inserted central catheter (PICC) or arteriovenous fistula;
* Presence of implanted cardiac devices, such as pacemakers, defibrillators, or cardiac resynchronization devices, which prevent ECG acquisition via smartwatch;
* Diagnosis of conditions associated with narrowing or obstruction of the aorta and subclavian arteries (e.g., Stanford Type A chronic aortic dissection, Takayasu arteritis, Subclavian Steal Syndrome, or Kawasaki disease), which may cause discrepancies in blood pressure between upper limbs and interfere with study assessments.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and number of Atrial Fibrillation (AF) events detected | During the monitoring period for each group, as specified (14-45 days depending on group)
  Incidence and total number of AF events detected, stratified by study group and device type (smartwatch, portable Holter). This allows assessment of AF detection rate across different monitoring protocols and devices during the follow-up period.
Number of critical health alerts generated by the FAPO-SI³ platform | During the monitoring period for each group, as specified (14-45 days depending on group)
  Alerts categorized by physiological parameter: blood pressure (BP), heart rate (HR), and oxygen saturation (SpO₂). Mean clinical response time to alerts will be calculated per patient during their respective monitoring period, allowing assessment of platform responsiveness and clinical workflow efficiency.
Patient risk classification generated by the AI model | During the monitoring period for each group, as specified (14-45 days depending on group)
  Distribution of patients across AI-generated risk categories (e.g., low, moderate, high) based on physiological and biometric data collected from the smartwatch and portable Holter system during the monitoring period.

SECONDARY OUTCOMES:
Patient risk classification generated by the AI model | During the monitoring period for each group, as specified (14-45 days depending on group)
  Distribution of patients across AI-generated risk categories adapted from the Manchester Triage System. The algorithm will classify patients into risk levels (e.g., immediate, very urgent, urgent, standard, non-urgent) based on physiological and biometric data collected from the smartwatch and portable Holter system during the monitoring period.
Adverse events related to device use | From enrollment through the monitoring period, up to 45 days depending on study group
  Incidence of device-related adverse events including skin lesions (MARSI), allergic reactions, and discomfort (graded using validated scales) reported during the monitoring period.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coracao, HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Participant monitoring will be conducted by the multidisciplinary team via the SI³ platform, allowing near real-time detection of clinical events and prompt intervention. After study completion, all data will be anonymized and analyzed by the InCor team. De-identified datasets may be shared with the sponsor and affiliated entities. No personally identifiable information will be disclosed. All data sharing will comply with ethical and legal data protection standards.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual participant data (IPD) and supporting documentation will be made available exclusively to the study sponsor following the completion of the clinical study. There is no defined end date, as the sponsor will assume full custodianship of the data upon transfer. No public sharing of the data is planned.
Access Criteria: Access to IPD and supporting information will be restricted to the study sponsor, in accordance with contractual agreements and applicable data protection regulations. The sponsor will have full authority over data access, management, and potential secondary use.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT07174206/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT07174206/ICF_001.pdf